CLINICAL TRIAL: NCT01490463
Title: Brain Lesions Following Endovascular and Surgical Treatment of Unruptured Intracranial Aneurysms: Incidence and Influence on Clinical Outcome in a Prospective Study.
Brief Title: Brain Lesions Following Endovascular and Surgical Treatment of Unruptured Intracranial Aneurysms
Acronym: LESUIA
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Department of Neurosurgery, Goethe-University Frankfurt am Main (Unknown); Institute of Neuroradiology, Goethe-University Frankfurt am Main (Unknown)
Responsible Party: Principal Investigator, Erdem Güresir, Department of Neurosurgery, Goethe-University Frankfurt am Main, Johann Wolfgang Goethe University Hospital
Other Study IDs: JohannWGUH_LESUIA
Record Dates: First submitted 2011-12-12; First posted 2011-12-13 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Unruptured Intracranial Aneurysms
Keywords: Treatment of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the incidence and impact of brain lesions in MRI after coiling and clipping of unruptured intracranial aneurysms on clinical and neurological outcome of patients.

DETAILED DESCRIPTION:
Silent ischemic lesions after treatment of unruptured intracranial aneurysm (UIA) might alter patients' clinical and neurological outcome. Furthermore silent brain lesions are not well documented after endovascular and surgical treatment of unruptured intracranial aneurysms. Therefore, the investigators investigate the incidence and influence of treatment-related ischemic lesions in magnetic resonance / diffusion-weighted-imaging after endovascular and surgical treatment of UIA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis and treatment of unruptured intracranial aneurysm
* age ≥ 18 yrs
* written informed consent by patients prior to study participation
* willingness to participate in follow-up

Exclusion Criteria:

* ruptured intracranial aneurysm
* contraindication for MRI
* Participation in an intervention-/AMG-study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unruptured intracranial aneurysm undergoing endovascular or surgical treatment
Sampling Method: Non-Probability Sample
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Platz J, Wagner M, Guresir E, You SJ, Konczalla J, de Rochemont RD, Berkefeld J, Seifert V. Early diffusion-weighted MRI lesions after treatment of unruptured intracranial aneurysms: a prospective study. J Neurosurg. 2017 Apr;126(4):1070-1078. doi: 10.3171/2016.2.JNS152456. Epub 2016 May 20. PMID 27203140